CLINICAL TRIAL: NCT03075592
Title: Post-ERCP Pancreatitis Severity Indication (PEPSI) Study
Acronym: PEPSI
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Georgios Papachristou, Professor of Medicine, University of Pittsburgh
Other Study IDs: IRB0609028
Record Dates: First submitted 2017-02-02; First posted 2017-03-09 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participant samples will be stored for an indefinite period of time in the Genomics and Proteomics Core Laboratories or in the laboratory of Dr. Whitcomb or appropriate core facility at the University of Pittsburgh. The samples will remain within the research studies of Dr. Whitcomb. Only authorized samples will be made available to other studies following IRB guidelines. The primary investigator, Dr. David Whitcomb, will have control over the blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERCP candidates: ERCP candidates

SUMMARY:
This study plans to directly address the problem of post-ERCP pancreatitis to gauge the various factors involved in its development and genetic variability in the immune response to an isolated pancreatic insult. In addition, the investigators hope to study markers of the early immune response to this injury and to develop a risk-assessment model.

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreaticography (ERCP) is an important diagnostic and therapeutic tool in the management of pancreatic and biliary diseases. However, it carries up to 10% risk of developing acute pancreatitis, 10% of which will be severe. Current models to predict the severity of acute pancreatitis are incomplete and unable to prognosticate early in the course of the disease because they are based on biomarkers of late immune response. Recent findings suggest that polymorphisms in the gene coding for MCP-1 (Monocyte Chemotactic Protein-1) play an important role in the early immune response leading to either mild versus severe acute pancreatitis of various etiologies.

This study plans to directly address the problem of post-ERCP pancreatitis to gauge the various factors involved in its development and genetic variability in the immune response to an isolated pancreatic insult. In addition, we hope to study markers of the early immune response to this injury and to develop a risk-assessment model.

ELIGIBILITY:
Inclusion Criteria:

1. All people presenting for ERCP procedures.
2. Males and females of 14 years of age and older.
3. Willingness to participate in the study and sign the informed consent. (Children will require a representative to sign the informed consent).
4. People in whom therapeutic pancreatic interventions are planned during the ERCP procedure.
5. Intact papilla

Exclusion Criteria:

1. Persons unwilling to sign the informed consent
2. Disorientation secondary to irreversible organic brain damage.
3. Hemoglobin of less than 11 gm/dl in children of 10 years of age to puberty and hemoglobin of 12 gm/dl in pubertal males and females.
4. Mean corpuscular volume (MCV) of less than 77 in all children of 18 years or younger.
5. ERCP scheduled for stent change
6. Previous diagnosis of pancreatic cancer or cholangiocarcinoma
7. History of chronic pancreatitis
8. Active Acute Pancreatitis prior to ERCP (typical pain and amylase or lipase >3 times UNL)or smoldering pancreatitis
9. History of Recurrent Acute Pancreatitis with chronic pain between acute attacks of >5/10 more than 3 days per week.
10. Previous sphincterotomy
11. Post surgical anatomy
12. History of organ transplant
13. On medications for the treatment of HIV

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 14 years of age and older, ERCP candidates.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop post ERCP pancreatitis as assessed by their clinical course | 1 year
  Develop a multi-factorial mathematical risk model that will help predict the exact risk for pancreatitis-associated complications of ERCP and to help power and structure future interventional studies.

SECONDARY OUTCOMES:
Number of patients with high serum amylase and cytokine levels as assessed by their clinical data. | 1 year
  Determine the relationship between pre and post-ERCP serum amylase and cytokine levels including IL-6, IL-8, CRP and MCP-1 and other injury or inflammatory markers as biomarkers of genetic polymorphisms in the corresponding genes.
Genetic markers that cause patients to develop post ERCP pancreatitis as identified by their genes | 1 year
  Determine if genetic polymorphisms of Monocyte Chemotactic Protein-1 (MCP-1) confer an increased risk for post-ERCP (Endoscopic Retrograde Cholangio- Pancreaticography) acute pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios I Papachristou, MD, Study Chair — Ohio State University